CLINICAL TRIAL: NCT06455462
Title: Patient Characteristics, Treatment Patterns and Outcomes of Patients With Severe Asthma Treated With Tezepelumab in the Real World; a Retrospective, Observational Medical Chart Review Conducted in UK Severe Asthma Centres
Acronym: TRAILBLAZE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5180R00027
Record Dates: First submitted 2024-03-01; First posted 2024-06-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Tezepelumab — tezepelumab treatment initiated between 1st January 2023 and 31st March 2024

SUMMARY:
This is a retrospective, observational chart review that will include patients with severe asthma (SA) who have participated in the tezepelumab patient access programme (TPAP). Electronic case report forms (eCRFs) will be used for data abstraction of clinical information from the health records of patients enrolled in the TPAP from up to eleven NHS trusts.

Approximately 350 patients with an index date (defined as the date of administration of the first dose of tezepelumab) between 1st January 2023 and 19th July 2023 (patients enrolled in the patient access programme), and between 20th July 2023 and 31st March 2024 (patients receiving tezepelumab in routine care), and meet the study eligibility criteria will be included in the study.

Participation in the study does not affect the patients' treatment decisions since all data will be collected retrospectively from medical records. Key study definitions include:

* Index date - the date of tezepelumab initiation (i.e., the date of first dose).
* Pre-index period - defined as any time prior to tezepelumab initiation
* Baseline period - defined as the 52 weeks prior to the index date
* Outcomes period - defined as the 52 weeks post-index date.

Patients will be followed up from their index date until the first of the following events (whichever is first): reach 52 weeks post-index, they switch to a different biologic treatment, die, or are otherwise lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received their first dose of tezepelumab between 1st January 2023 and 19th July 2023 (TPAP cohort) or between 20th July 2023 and 31st March 2024 (post-TPAP cohort)
* Patients aged ≥18 years at index

Exclusion Criteria:

* Patients who received any biologic drug for the treatment of asthma in a clinical trial at any time during the 52 weeks prior to the index date.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SA treated with tezepelumab as part of the TPAP (who received their first dose between 1st January 2023 and 19th July 2023) or post-TPAP (between 20th July 2023 and 31st March 2024) will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Annualised exacerbation rate | 24 weeks, 52 weeks

SECONDARY OUTCOMES:
Exacerbation rate during the baseline | Baseline (-52 to 0 weeks)
Change from baseline in annual exacerbation rate | Baseline (-52 to 0 weeks) to 52 weeks
  Absolute and relative change will be described
Exacerbation rate by season | 52 weeks
Time to first exacerbation | 52 weeks
Proportion of patients recieving maintenance oral corticosteroids (mOCS) for asthma (y/n) | Baseline (-52 to 0 weeks), after 24 and 52 weeks
Dose of mOCS for asthma | Baseline (-52 to 0 weeks), after 24 and 52 weeks
Change from baseline in dose of mOCS for asthma | Baseline (-52 to 0 weeks), after 24 and 52 weeks
  Absolute and relative change will be described
Summary measures of Asthma Control Questionnaire (ACQ-6) score | Baseline (-52 to 0 weeks), after 24 and 52 weeks
Change since baseline in ACQ-6 score | Baseline (-52 to 0 weeks) to 52 weeks
  Absolute and relative change will be described
Proportion achieving MCID change in ACQ-6 | 52 weeks
Proportion achieving 2xMCID change in ACQ-6 | 52 weeks
Quality of life measured by the Asthma Quality of Life Questionnaire (AQLQ) | Baseline (-52 to 0 weeks), after 24 and 52 weeks
  AQLQ-12 or mini-AQLQ will be measured separately.
Change from baseline in AQLQ score | Baseline (-52 to 0 weeks) to 52 weeks
  Absolute and relative change will be described
Proportion achieving MCID change in AQLQ | 52 weeks
Proportion achieving 2xMCID change in AQLQ | 52 weeks
Summary measures of forced expiratory volume in 1 second (FEV1) | Baseline (-52 to 0 weeks), after 24 and 52 weeks
Change from baseline in FEV1 | Baseline (-52 to 0 weeks) and 52 weeks
  Absolute and relative change will be described
Summary measures of % predicted FEV1 | Baseline (-52 to 0 weeks), after 24 and 52 weeks
Summary measures of FEV1/FVC | Baseline (-52 to 0 weeks), after 24 and 52 weeks
Summary measures of fractional exhaled nitric oxide (FeNO, ppb) | Baseline (-52 to 0 weeks), after 24 and 52 weeks
Change from baseline in FeNO | Baseline (-52 to 0 weeks) and 52 weeks
  Absolute and relative change will be described
Hightest FeNO level (ppb) recorded in patient record | Any time prior to tezepelumab initiation
Summary measures of blood eosinophil count | Baseline (-52 to 0 weeks), after 24 and 52 weeks
Change from baseline in blood eosinophil count (BEC) | Baseline (-52 to 0 weeks) and 52 weeks
  Absolute and relative change will be described
Hightest blood eosinophil count recorded in patient record | Any time prior to tezepelumab initiation
Summary measures of IgE | Baseline (-52 to 0 weeks), after 24 and 52 weeks
Change from baseline in IgE | Baseline (-52 to 0 weeks) and 52 weeks
  Absolute and relative change will be described
Hightest IgE level recorded in patient record | Any time prior to tezepelumab initiation
Proportion of patients recieving treatment with LABA, LAMA or ICS | Baseline (-52 to 0 weeks), 24 weeks and 52 weeks
  Asthma related treatment with LABA, LAMA and/or ICS will be described
Summary measures of inhaled corticosteroid (ICS) dose | Baseline (-52 to 0 weeks), after 24 and 52 weeks
  Asthma-related ICS use will be described
Proportion of patients with previous biologic use | Baseline (-52 to 0 weeks)
Number of previous biologics prior to tezepelumab initiation | Any time prior to tezepelumab initiation
Reason for tezepelumab initiation | Baseline (-52 to 0 weeks)
Time to tezepelumab discontinuation | Baseline (-52 to 0 weeks) to 52 weeks
Number, type and rate of asthma related hospitalisation events | Baseline (-52 to 0 weeks) to 52 weeks
Number and rate of asthma related A&E visits | Baseline (-52 to 0 weeks) to 52 weeks
Number and rate of asthma related ICU admissions | Baseline (-52 to 0 weeks) to 52 weeks
Number and rate of asthma related ventilator use | Baseline (-52 to 0 weeks) to 52 weeks
Number and rate of asthma related outpatient visits | Baseline (-52 to 0 weeks) to 52 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - Research Site, Birmingham
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Newcastle
  - Research Site, Plymouth
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/